CLINICAL TRIAL: NCT03545477
Title: Assessment of the Rehabilitative Effects of Curved-walking Training in Stroke, Parkinson and Orthopaedic Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Dept. of Electronics, Informatics, Bioengineering, Politecnico di Milano, Italy (Other)
Responsible Party: Principal Investigator, Giorgio Ferriero, Scientific Director, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2152CE
Record Dates: First submitted 2018-04-24; First posted 2018-06-04 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Stroke, Acute; Parkinson Disease; Femur Fracture
Keywords: gait rehabilitation; curved walking training; lower limb
MeSH Terms: conditions — Stroke; Parkinson Disease; Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel treatment, curved-walking training (Experimental): It consists of 20 sessions of training (three times a week for seven weeks) composed by standard physical therapy and a novel approach to locomotion rehabilitation based on curved-walking training. Each session lasts about 90 minutes.
  Interventions: Other: Novel locomotion treatment: curved-walking training; Other: Standard physical therapy
- Usual care (Active Comparator): It consists of 20 sessions of training (three times a week for seven weeks) of standard physical therapy and conventional straight-walking training. Each session lasts about 90 minutes.
  Interventions: Other: Standard locomotion treatment: straight-walking training; Other: Standard physical therapy

INTERVENTIONS:
Other: Novel locomotion treatment: curved-walking training — Each training session is comprehensive of a 30-minute walking training on curved trajectory ("S" trajectory composed by two semicircle with a radius of 1.2 m)
  Arms: Novel treatment, curved-walking training
Other: Standard locomotion treatment: straight-walking training — It consists of 30 minutes of locomotion training on straight trajectories, as typically proposed during traditional gait rehabilitation
  Arms: Usual care
Other: Standard physical therapy — It consists of 60 minutes of stretching, muscular conditioning and coordination,postural exercises for trunk control, standing, functional exercies and upper limb rehabilitation, customized on patient's need.

SUMMARY:
The recovery of walking ability is crucial to promote independence in daily living and is one of the major goal of neuromotor rehabilitation.

Currently, standard rehabilitative programs are usually based on straight-walking training (SWT) and the assessment of their effects is performed through functional scales based on straight-walking trajectories, e.g. Timed Up and Go (TUG), 10 meters walking test (10mWT).

Curved-walking training (CWT) may be interesting to provide an ecological and challenging context during rehabilitation. Indeed, CWT is based on demanding neural processes that drive an asymmetrical contribution at lower limb level, challenging balance ability and complex adaptation such as body weight shifting in response to centrifugal force and production of different step lengths.

Up to now, literature has investigated CWT in healthy adults in terms of muscular activation, kinematics and kinetics of the movement. Results showed that CWT needs a different biomechanical strategy with respect to SWT. Nevertheless CWT has not been investigated in pathological adults.

The present study aims at assessing the effectiveness of a rehabilitative physical therapy based on CWT with respect to traditional SWT for the recovery of locomotor abilities in neurological and orthopaedic patients.

The hypothesis is that a training based on curved-walking is ecologically meaningful and may be superior with respect to standard training in improving balance, walking abilities, and independence in activity of daily live of patients.

A secondary aim of the project is to propose an innovative functional scale based on the timed up and go on curved trajectory (CTUG), and to determine its reliability and responsiveness, establishing the minimum Detectable Change (MDC) and the Minimal Clinically Important Difference (MCID).

A single-blind randomized controlled study is being carried out on three different populations:

* Post-acute stroke patients
* Idiopathic Parkinson Disease
* Femoral fracture

A healthy group is also being recruited to provide reference values of CTUG. For each of the three populations, subjects are randomized into two groups. The experimental one performs a novel rehabilitative program composed by a 30-minute training on curved trajectory ("S" trajectory composed by two semicircle with a radius of 1.2 m) in addition to usual care. The control group performs an equal dose of traditional treatment on straight trajectories.

Both groups undergo 20 90-minutes sessions of training (three times a week for seven weeks).

Participants are evaluated at baseline (T0), after training (T1), and at a three-months follow-up visit (T2).

The primary outcome measure is the 10mWT (minimal clinically important difference of 0.16 m/s identified by Tilson and colleagues). On the basis of this measure, a sample size of 70 subjects for each population was computed.

ELIGIBILITY:
Inclusion Criteria:

* Post-acute stroke patients experiencing a stroke less than 6 months before recruitment
* Idiopathic Parkinson Disease with disability level from moderate to severe (modified Hoehn & Yahr scale 2.5-4)
* Femoral fracture, less than 1 month form surgery

Exclusion Criteria:

* Cognitive deficits (Mini Mental Scale Evaluation < 24)
* Hemineglect
* Modified Ashworth Scale of lower limb >2
* Unstable pharmacological treatment for Parkinson's Disease during the 15 days before the recruitment
* cardiopathic conditions
* metabolic conditions (e.g. dialysis) that prevent patients from aerobic training
* Previous history of major neurological, vascular, musculoskeletal disorders
* Body Mass Index > 30 Kg/m2
* Invasive pharmacological treatment or surgery for Parkinson's disease
* lower limb pain (VAS >3)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in 10 meter walk test (10MWT) | Baseline, 7 weeks, 20 weeks
  Time (seconds) needed by patients to walk for 10 meters

SECONDARY OUTCOMES:
curved-walking test | Baseline, 7 weeks, 20 weeks
  Time (seconds) needed to complete the "S" curved trajectory (7.53 m)
Timed Up and Go (TUG) | Baseline, 7 weeks, 20 weeks
  Time (seconds) needed to the patient to stand up upon therapist's command, walk 3 meters, turn around, walk back to the chair and sit down.
Curved Timed Up and Go | Baseline (test), day 2 (retest), 7 weeks, 20 weeks
  Time (seconds) needed to the patient to stand up upon therapist's command, walk 3 meters following the curved trajectory, turn around, walk back on the curved trajectory to the chair and sit down.
Balance test | Baseline, 7 weeks, 20 weeks
  Balance performance assessed by Balance test. Postural stability is evaluated using the commercial balance board Balance Master basicTM, NeuroCom® International, Inc. Assessments evaluate the postural sways during upright stance both with eyes open and closed; the limits of stability in different directions (forward, backward, right, and left); and the capability to shift the weight both left/right and forward/backward.
Pain Numerical Rating Scale | Baseline, 7 weeks, 20 weeks
  Pain perceived on 11 levels (0-10)
Short Form Healthy Survey SF-36 | Baseline, 7 weeks, 20 weeks
  Healthy status investigated in 36 questions
Falls Efficacy Scale (FES) | Baseline, 7 weeks, 20 weeks
  Risk of falls evaluated with 10 elements, each scored from 0 to 10. A total score higher than 70 suggests fear of falls.
Global Perceived Effect (GPE) for patients | 7 weeks
  Perceived effectiveness of training for patients. A score from 1 (significantly improved) to 7 (significantly worsened) is assigned.
Global Perceived Effect (GPE) for physiotherapists | 7 weeks
  Perceived effectiveness of training for physiotherapists. A score from 1 (significantly improved) to 7 (significantly worsened) is assigned.
Motricity Index (MI) | Baseline, 7 weeks, 20 weeks
  Functional ability of limb - post-stroke population only. The quality of different limb movement are scored from 0 to 33 points, with a total score of 100 for each limb
39-Item Parkinson's Disease Questionnaire (PDQ-39) | Baseline, 7 weeks, 20 weeks
  Quality of life questionnaire - Parkinson's Disease only. The questionnaire is based on 39 questions and the total score ranges from 0% (no difficulty) to 100% (maximum level of difficulty)
Tampa Scale for Kinesiophobia (TSK) | Baseline, 7 weeks, 20 weeks
  Fear of movement - Parkinson's Disease only. Score ranges from 13 (no fear) to 52 (maximum fear).
Unified parkinson's Disease Rating Scale (UPDRS) | Baseline, 7 weeks, 20 weeks
  Parkinson's Disease prognosis information - Parkinson's Disease only. Score ranges from 0 (normal) to 199 (severe impairment).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 7 weeks, 20 weeks
  Physical functionality, pain and stiffness - post-femoral fracture only. Its score ranges from 0 (high healthy status) to 100 (low healthy status)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Ferriero, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri Spa, Scientific institute of Lissone
Locations (1):
- Istituti Clinici Scientifici Maugeri Spa, Scientific Institute of Lissone, Lissone, Monza E Brianza, Italy

REFERENCES:
- [Background] Tilson JK, Sullivan KJ, Cen SY, Rose DK, Koradia CH, Azen SP, Duncan PW; Locomotor Experience Applied Post Stroke (LEAPS) Investigative Team. Meaningful gait speed improvement during the first 60 days poststroke: minimal clinically important difference. Phys Ther. 2010 Feb;90(2):196-208. doi: 10.2522/ptj.20090079. Epub 2009 Dec 18. PMID 20022995
- [Background] Courtine G, Papaxanthis C, Schieppati M. Coordinated modulation of locomotor muscle synergies constructs straight-ahead and curvilinear walking in humans. Exp Brain Res. 2006 Apr;170(3):320-35. doi: 10.1007/s00221-005-0215-7. Epub 2005 Nov 19. PMID 16328271
- [Background] Courtine G, Schieppati M. Human walking along a curved path. I. Body trajectory, segment orientation and the effect of vision. Eur J Neurosci. 2003 Jul;18(1):177-90. doi: 10.1046/j.1460-9568.2003.02736.x. PMID 12859351
- [Background] Godi M, Turcato AM, Schieppati M, Nardone A. Test-retest reliability of an insole plantar pressure system to assess gait along linear and curved trajectories. J Neuroeng Rehabil. 2014 Jun 5;11:95. doi: 10.1186/1743-0003-11-95. PMID 24903003